CLINICAL TRIAL: NCT04732234
Title: Pre-emptive Ultrasound Guided Superior Hypogastric Plexus Block in Pelvic Cancer Surgeries : a Randomized Double-Blinded Study
Brief Title: Pre-emptive US Guided Superior Hypogastric Plexus Block in Pelvic Cancer Surgeries : a Randomized Double-Blinded Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Abdelfattah Abdelwadod, Mohammed Abdelfattah Abdelwadod, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORG0003381-AP2006-50103
Record Dates: First submitted 2020-12-25; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Group S (SHPB group 18 ultrasound guided SHPB ) using 20 ml Bupivacaine 0.5% before skin incision.
  Group C (Control group 18 patients) in which same technique will be done but using normal saline 0.9%
Who Masked: Participant, Investigator
Masking Description: Randomization is done using computer generated sequence. Concealment will be achieved by opaque envelope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ( Group A) (Active Comparator): ultrasound guided superior hypogastric plexus block using 20 ml Bupivacaine 0.5% before skin incision.
  Interventions: Procedure: Superior Hypogastric Plexus Block
- (Group B) (Placebo Comparator): ultrasound guided superior hypogastric plexus block using 20 ml normal saline 0.9% instead of bupivacaine.
  Interventions: Procedure: Superior Hypogastric Plexus Block

INTERVENTIONS:
Procedure: Superior Hypogastric Plexus Block — Pre operative ultrasound guided superior hypogastric plexus block in pelvic surgeries using a curvilinear probe below umbalicus with needle in plane technique to reach the plexus in front of L5 vertebra

SUMMARY:
The superior hypogastric plexus (SHP) is a retroperitoneal structure with a predominance of afferent sympathetic nerve fibers. The perception of central pelvic pain is thought mainly to involve transmission through this plexus. Therefore, blocking or of SHP has been used to treat pelvic pain.

DETAILED DESCRIPTION:
Ultrasound guided superior hypogastric plexus block there is 2 equal groups:

Group S (SHPB group 18 patients) ultrasound guided SHPB is done after induction of balanced general anesthesia (fentanyl, propofol and rocuronium) using 20 ml Bupivacaine 0.5% before skin incision, Group C (Control group 18 patients) in which same technique will be done but using normal saline 0.9% instead of bupivacaine. Patients of both groups will receive patient controlled analgesia using morphine with continous background infusion of morphine 1.5 mg/h with adding granisterone 2mg/60 ml and ability to give bolus of 0.5 mg morphine on demand.

• Dosing and administration; Group S (SHPB group 18 ultrasound guided SHPB ) using 20 ml Bupivacaine 0.5% before skin incision.

Group C (Control group 18 patients) in which same technique will be done but using normal saline 0.9%

ELIGIBILITY:
Inclusion Criteria:

* ASA II,III.
* Patients undergoing pelvic surgeries.

Exclusion Criteria:

* Patients refusal,
* Coagulopathy,
* Infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | baseline till 24 hours postoperative
  Total 24 hours morphine consumption in milligrams

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | Visual analogue scale (VAS) at baseline till 24 hours postoperative
  scale in which 0 is least pain and 10 is sever pain

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed abdel wadod, MD, Principal Investigator — Anesthesia & pain management Dept, National Cancer Institute-Cairo - Egypt
Locations (1):
- Nataional Cancer Instituite, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided